CLINICAL TRIAL: NCT03137511
Title: Optimizing Access to Care Through New Technologies: a Randomized Study Evaluating the Impact of Telephone Contact and the Sending by the General Practitioner of Suspicious Lesions Melanoma Photographs Taken With a Smartphone, on the Time Limit to the Consultation With a Dermatologist
Acronym: OASE Melanome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RC16_0033
Record Dates: First submitted 2017-04-28; First posted 2017-05-02 (Actual); Last update posted 2019-04-29 (Actual); Status verified 2019-04

CONDITIONS: Patients at Risk for Melanoma
Keywords: Public Health; General Medicine; Dermatology

STUDY DESIGN:
Intervention Model Description: Cluster randomization of MGs corresponding to their exercise sites
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): General practitioners will be invited to screen for melanoma as part of their regular consultations.
  * The MG collects relevant clinical information
  * The MG takes 2 photographs of the lesion with his smartphone.
  * The MG sends to the dermatologist by e-mail the 2 photographs of the lesion accompanied by relevant clinical information
  * The MG calls the secretariat of the dermatologist to record the admissibility of the mail, to give the identity and the coordinates of the patient whose photos have just been sent and to obtain an appointment.
  * The dermatologist proposes an appointment to the patient.
  Interventions: Other: Taking photographs of suspicious lesions with his smartphone and sending them to the dermatologist
- Control group (No Intervention): General practitioners will be invited to screen for melanoma as part of their regular consultations.
  General practitioners and dermatologists continue their practice in the usual way.

INTERVENTIONS:
Other: Taking photographs of suspicious lesions with his smartphone and sending them to the dermatologist — Taking photographs of suspicious lesions with his smartphone and sending them to the dermatologist
  Arms: Intervention group

SUMMARY:
Early detection of melanoma showed an impact on the thickness of the lesions at the time of diagnosis. One challenge is to improve the modalities.

Decrease the rate of non-compliant patients among patients referred to the dermatologist for a suspicious lesion (patients who will never go to the consultation), and reduce the time interval between the first identification of the lesion and the excision allowing the diagnosis are major issues.

Direct contact between the general practitioner (GP) and the dermatologist would probably make it possible to shorten the care pathway of patients with lesions justifying excision.

The objective is to evaluate whether contacting the dermatologist directly by telephone and e-mailing the photograph of a suspicious melanoma lesion can significantly reduce the time required for access to the consultation for the following patients: (a) referred for a suspicious lesion of melanoma by the GP (b) and having a sufficiently suspicious lesion of melanoma so that the dermatologist conclude at the need for excision (true positives).

Expected results: The procedure should shorten the care pathway for patients with melanoma and decrease the proportion of patients who do not consult the dermatologist when they were referred ("non-observing patients").

This should facilitate the identification of thinner lesions. The benefit for the patient is then direct with a survival at 5 years higher.

In public health terms, it is expected a benefit as better optimization of resources. In a situation of shortage of professionals, access to the dermatologist should be optimized by optimizing emergency access for patients who require it.

ELIGIBILITY:
Inclusion Criteria:

Patients:

* Consulting a general practitioner participating in the study,
* Having a suspicious cutaneous lesion of melanoma according to the MG,
* Referred to a dermatologist who agreed to participate in the study,
* > = 18 years of age, with written informed consent,
* Affiliated to a social security scheme

Exclusion Criteria:

Patients:

* Consulting a general practitioner who does not participate in the study,
* Having no suspect melanoma lesion according to MG,
* Referred to the dermatologist for symptoms or pathologies unrelated to a suspicion of melanoma
* Wishing to consult a dermatologist who refused to participate in the study,
* Refusing the transmission by mail of 2 anonymised photos,
* <18 years of age, or with no written informed consent.
* Major under tutelage, under curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 270 (Actual)
Dates: Start 2017-05-23 (Actual); Primary Completion 2018-11-28 (Actual); Study Completion 2018-11-28 (Actual)

PRIMARY OUTCOMES:
Time limit for consultation general practitioner / dermatologist, patients having a sufficiently suspicious lesion of melanoma | 12 months
  Time limit for consultation between consultation of the general practitioner and consultation with the dermatologist, for patients:
  1. referred for a suspicious lesion of melanoma by the general practitioner,
  2. and having a sufficiently suspicious lesion of melanoma so that the dermatologist conclude at the need for excision

SECONDARY OUTCOMES:
Time limit for consultation general practitioner / dermatologist, patients NOT having a sufficiently suspicious lesion of melanoma | 12 months
  Time limit for consultation between consultation of the general practitioner and consultation with the dermatologist, for patients:
  1. referred for a suspicious lesion of melanoma by the general practitioner,
  2. BUT NOT having a sufficiently suspicious lesion of melanoma so that the dermatologist conclude at the need for excision
"Non-observing" patients between the 2 randomization groups | 12 months
  Proportion of "non-observing" patients between the 2 randomization groups. A non-observing patient is a patient who has not consulted a dermatologist within 12 months following the prescription of his or her GP.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, Nantes, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bouton C, Schmeltz H, Leveque C, Gaultier A, Quereux G, Dreno B, Nguyen JM, Rat C. Early diagnosis of melanoma: a randomized trial assessing the impact of the transmission of photographs taken with a smartphone from the general practitioner to the dermatologist on the time to dermatological consultation. BMC Health Serv Res. 2024 May 24;24(1):660. doi: 10.1186/s12913-024-11106-9. PMID 38783296